CLINICAL TRIAL: NCT00215293
Title: A Randomized Multi-Center Study to Evaluate the Safety and Efficacy of the Cervical I/F Cage for Anterior Cervical Fusion
Brief Title: Cervical I/F Cage for Anterior Cervical Fusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G000019
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Cervical Intervertebral Disc Degeneration
Keywords: fusion; cervical; spine
MeSH Terms: interventions — Transplantation, Autologous; Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical Cage (Experimental): Cervical I/F Cage
  Interventions: Device: Cervical I/F Cage
- Graft Spacer (Active Comparator): Autograft or allograft with a plate, or autograft alone.
  Interventions: Device: Autograft or allograft with a plate, or autograft alone.

INTERVENTIONS:
Device: Cervical I/F Cage
  Arms: Cervical Cage
Device: Autograft or allograft with a plate, or autograft alone.
  Arms: Graft Spacer

SUMMARY:
The purpose of this study is to determine the clinical success of the Cervical I/F Cage in treatment of one or two adjacent levels of degenerative disc disease of the cervical spine compared with standard of care treatment using either autograft, autograft with a plate or allograft with a plate

DETAILED DESCRIPTION:
This is a prospective randomized multi-center clinical trial to assess the safety and efficacy of the investigational device, Cervical I/F Cage for fusion in one or two adjacent levels of the cervical spine. Patients will be randomly assigned in a ration of 1:1 between the investigational and control groups.

Comparison: The device will be compared to a control group consisting of the 3 accepted standard of care treatments (autograft, autograft with an anterior plate, or allograft with an anterior plate). For two level fusions, the control group will be limited to autograft with a plate or allograft with a plate. Based on the current literature, it is believed that there is no difference between the three treatments in terms of clinical success, fusion success, or safety issues. However, amongst the investigators there are preferred treatments. Each investigator will choose one or more of the control treatments at study initiation. Patients will then be randomized in a 1:1 Cage:control randomization schema. Approximately 240 subjects will be enrolled at 20 sites. Eligible patients will have symptomatic degeneration of one or two adjacent cervical discs, have failed six weeks of non-surgical treatment, have sufficiently severe enough symptoms to warrant surgery, and have had no prior fusion surgery on the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Persistent recurrent neck and/or shoulder and arm pain refractory to 6 weeks of non-surgical therapy.
* Radiographic evidence of significant disc degeneration at one or two adjacent cervical levels (C4-7)

Exclusion Criteria:

* Significant degeneration at more than two cervical levels,
* Prior surgical treatment of the cervical spine; laminotomy or foraminotomy allowed,
* Gross instability due to trauma,
* Disability in the lumbar spine,
* Infection in the disc or spine, past or present,
* Any active infection at time of surgery,
* Tumor in the spine,
* Significant osteoporosis or metabolic bone disease,
* Pregnant, lactating or wishes to become pregnant within duration of the study,
* Refusal to accept the use of autograft tissue.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2000-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Fusion Status | 24 months
Neck Disability Index
Neurological Status
Secondary Surgical Interventions

SECONDARY OUTCOMES:
Adverse Events
Donor Site Pain
Neck Pain
Arm Pain
Disc Space Height
Sagittal Alignment
SF-36, Health Related Quality of Life